CLINICAL TRIAL: NCT03826849
Title: A Pilot Evaluation of the Insomnia Coach Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Kuhn, Clinical Psychologist, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-47188
Record Dates: First submitted 2019-01-04; First posted 2019-02-01 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Insomnia; Trauma, Psychological
Keywords: mobile app; Veteran; cognitive behavioral therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): Assessment only condition for all 12 weeks of participation.
- Insomnia Coach (Experimental): Intervention condition that involves use of the Insomnia Coach app for 6 weeks.
  Interventions: Behavioral: Insomnia Coach

INTERVENTIONS:
Behavioral: Insomnia Coach — Insomnia Coach is a mobile application that provides psychoeducation and self-management tools for insomnia symptoms based on cognitive behavioral therapy for insomnia (CBT-I)
  Arms: Insomnia Coach

SUMMARY:
This pilot study is designed to test the feasibility, acceptability, and potential effectiveness of a mobile phone application (app) developed by the VA National Center for PTSD (VA NCPTSD) for use by Veterans with insomnia. The primary objective is to assess whether Veterans find the Insomnia Coach app to be satisfactory and feasible to use. Secondary objectives are to determine if use of the app improves subjective sleep quality and sleep parameters (e.g., sleep latency, wake after sleep onset, and total sleep time), as well as other important outcomes (e.g., daily functioning).

DETAILED DESCRIPTION:
There are high rates of insomnia among Veterans, particularly those who have been exposed to potentially traumatic situations (i.e., combat exposure) and few receive cognitive-behavioral therapy for insomnia (CBT-I), a first-line treatment for insomnia. Insomnia Coach is a mobile app for individuals with insomnia symptoms. This app provides:

* education about sleep, the development of insomnia, and evidence based behavioral and cognitive strategies
* self-assessment tools measuring insomnia severity and sleep need
* self-monitoring with a daily sleep diary
* self-management tools for relaxation and changing thinking about sleep
* individualized recommendations for a preferable sleep window (i.e., bed and rise times)
* daily reminders for behavioral changes In this pilot randomized controlled trial (RCT), 50 Veterans with significant insomnia symptoms will be recruited using flyers and social media (i.e., Facebook ads) and randomized in equal numbers to receive one of two conditions: 1) the Insomnia Coach mobile app (which is based on cognitive-behavioral therapy for insomnia (CBT-I)) and, 2) a waitlist control.

Objective use of the Insomnia Coach mobile app will be tracked to assess feasibility (i.e., will participants use the app as intended). Participants will complete measures (using Qualtrics) of sleep, insomnia severity, depression and anxiety, and functional well-being at baseline, 6 weeks (posttreatment), and 12 weeks (follow-up). At post-treatment, participants in the Insomnia Coach app condition will also be asked to report their level of satisfaction with the app and to complete a brief qualitative evaluation of their experience using the app. Waitlist control condition participants will be informed about the Insomnia Coach app and provided with information on how to download it after completion of the follow-up assessment (i.e., at 12 weeks).

The aim of this research is to learn whether individuals, particularly Veterans, with insomnia, find Insomnia Coach to be satisfactory and feasible to use. It also aims to assess if use of the app potentially improves subjective sleep quality and sleep parameters (e.g., sleep latency, wake after sleep onset, and total sleep time), as well as other important outcomes (e.g., daily functioning). If this research demonstrates that Insomnia Coach is a promising tool for individuals experiencing sleep difficulties, it has the potential to address a need using a very cost-effective, widely accessible, scalable solution that would warrant more rigorous evaluation (e.g., a full-scale RCT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55
* Owner of smartphone or tablet with Android or iOS operating system
* Probable insomnia (i.e., ISI >=10, 3 months or more with sxs, occurring >= 3 days/week, 30 minutes or > with sleep loss)
* Able to read/write English
* Internet connection and active email address

Exclusion Criteria:

* Comorbid sleep disorders (apnea, RLS, narcolepsy)*
* Started or changed dosage of sleep medications or SSRIs in past 2 months
* Unstable housing
* Medical condition identifiably causing sleep problems
* Significant alcohol/drug use issues
* Current mania or psychosis
* Currently severely depressed (PHQ-9 >20)
* Currently receiving or having recently received insomnia therapy resembling CBT-I
* Shift working
* Pregnant
* Newborn (3 mos. or younger) living in residence
* < 5 hours of average total sleep time on 7 days of sleep diaries

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Objective App Usage Data | 6 weeks
  Composite of app usage data comprised of button taps, sections visited, self-entered data, number of visits and days used, and time spent on the app per visit. Various combinations and aggregations of these behaviors will be explored as best indicators to optimally summarize app use.
Mobile Apps Rating Scale (MARS; Stoyanov et al., 2015) | 6 weeks
  A 20-item multidimensional, objective measure of app usability. It includes four subscales that measure an app's engagement, functionality, aesthetics, and information quality. All items are rated on a 5-point scale from "1. Inadequate" to "5. Excellent". The scores are tallied up and a mean score out of 5 is given to each of the categories scored.
System Usability Scale (SUS; Brooke, 1986) | 6 weeks
  A 10-item questionnaire of usability of products and services, including hardware, software, mobile devices, websites and applications. Items are on a 5-point scale numbered 1 to 5. Half of the items are worded negatively and half are worded positively. SUS yields a single number representing a composite measure of the overall usability of the system. To calculate the SUS score, the score contributions from each item are summed. Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Then the sum of the scores is multiplied by 2.5 to obtain the overall value of SU. SUS scores have a range of 0 to 100.
Qualitative Interview (Kuhn & Miller, 2018) | 6 weeks
  A 24-question, semi-structured interview to assess users' perceptions of Insomnia Coach.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI; Bastien et al., 2011) | 6 and 12 weeks
  A 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia symptoms in the past month. Items are on a scale from 0 to 4. The seven answers are added up to get a total score, with higher scores reflecting greater insomnia severity
Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) | 6 and 12 weeks
  A 19-item self-report measure assessing qualities and problems associated with sleep in the past month. It generates seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. A global sleep quality score is obtained by summing the seven component scores. Higher scores reflect poorer sleep quality. The global score ranges from 0 to 21, with a cut-off score of 5 as distinguishing "good" sleepers from "poor" sleepers.
PROMIS-Sleep-Related Impairment (PROMIS-SRI; Buysse et al., 2010) | 6 and 12 weeks
  This 16-item self-report form assesses sleep-related impairment over the past seven days. Each question has five response options ranging in value from 1 to 5. To find the total raw score the values of the response to each question are summed. The raw scores are converted to a standardized T-score using conversion tables published on the PROMIS website (nihpromis.org), with higher scores indicating greater sleep/wake disturbances.
Consensus Sleep Diary: Change in sleep onset latency (Carney et al., 2012) | 6 and 12 weeks
  The Consensus Sleep Diary will be used to prospectively monitor self-reported sleep. Shorter sleep onset indicates faster time to fall asleep.
Consensus Sleep Diary: Change in wake after sleep onset (Carney et al., 2012) | 6 and 12 weeks
  The Consensus Sleep Diary will be used to prospectively monitor self-reported sleep. Less time spent awake during the sleep period indicates better sleep.
Consensus Sleep Diary: Change in sleep efficiency (Carney et al., 2012) | 6 and 12 weeks
  The Consensus Sleep Diary will be used to prospectively monitor self-reported sleep. Higher sleep efficiency (total sleep time/time spent in bed) indicates better sleep quality.
Generalized Anxiety Disorder - 7 Item (GAD-7; Spitzer et al., 2006) | 6 and 12 weeks
  This 7-item measure assesses anxiety symptom severity. Items are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Patient Health Questionnaire 8 (PHQ-8; Kroenke et al., 2009) | 6 and 12 weeks
  An 8-item self-report instrument used to assess depression severity. Since the scale is self-administered in our studies and further probing about positive responses is not feasible, the question about suicide from the PHQ-9 was removed. Items are scored 0 to 3, with the total score being the sum of the 8 items. Higher scores indicate greater depression severity, with a score of 10 or greater considered major depression, and scores of 20 or more is severe major depression.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No